CLINICAL TRIAL: NCT04680884
Title: Empirical Steroids and/or Antifungals in Immunocompromised Patients With Acute Respiratory Failure From Undetermined Etiology: a Multicenter Double-blind Randomized Controlled Trial
Acronym: EFRAIM II
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: APHP180584
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Acute Respiratory Failure; Immunocompromised Patients
MeSH Terms: interventions — Steroids; Antifungal Agents; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental for steroid (Experimental): 2 mg/kg/day of IV methylprednisolone for three days. As of day 4, the daily dose will be tapered to 1 mg/kg/day until day 7, followed by 0,5 mg/kg/day from day 8 to day 14 + IV placebo of isavuconazole
  Interventions: Drug: Experimental for steroid
- Experimental for antifungals (Experimental): IV placebo of methylprednisolone + IV isavuconazole (200 mg every 8 hours for 2 days followed by 200 mg per day until ICU discharge or for a total duration of 14 days)
  Interventions: Drug: Experimental for antifungals
- Experimental for steroids and antifungals (Experimental): IV methylprednisolone 2 mg/kg/day for three days. As of day 4, the daily dose will be tapered to 1 mg/kg/day until day 7, followed by 0.5 mg/kg/day from day 8 to day 14 + IV isavuconazole 200 mg every 8 hours for 2 days followed by 200 mg per day until ICU discharge or for a total duration of 14 days)
  Interventions: Drug: Experimental for steroids and antifungals
- Best standard of care (Other): IV placebo of methylprednisolone + IV placebo of isavuconazole. This group receives the treatment that is currently recommended.
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Experimental for steroid — 2 mg/kg/day of IV methylprednisolone for three days. As of day 4, the daily dose will be tapered to 1 mg/kg/day until day 7, followed by 0,5 mg/kg/day from day 8 to day 14 + IV placebo of isavuconazole
  Arms: Experimental for steroid
Drug: Experimental for antifungals — IV placebo of methylprednisolone + IV isavuconazole (200 mg every 8 hours for 2 days followed by 200 mg per day until ICU discharge or for a total duration of 14 days)
  Arms: Experimental for antifungals
Drug: Experimental for steroids and antifungals — IV methylprednisolone 2 mg/kg/day for three days. As of day 4, the daily dose will be tapered to 1 mg/kg/day until day 7, followed by 0.5 mg/kg/day from day 8 to day 14 + IV isavuconazole 200 mg every 8 hours for 2 days followed by 200 mg per day until ICU discharge or for a total duration of 14 days)
  Arms: Experimental for steroids and antifungals
Other: Standard of care — IV placebo of methylprednisolone + IV placebo of isavuconazole. This group receives the treatment that is currently recommended.
  Arms: Best standard of care

SUMMARY:
Acute respiratory failure (ARF) is the leading reason of ICU admission in immunocompromised patients. Failure to identify the ARF etiology is associated with increased mechanical ventilation and mortality rates. This was confirmed in the large Efraim 1 study published in 2017, where undetermined ARF etiology affected 609/1611 (38%) patients at day 3, 402 (25%) patients at day 7 and 199 (12.3%) patients overall, and was associated with a case fatality of 55% (vs. 40% in other patients). In lung biopsy/autopsy findings from these patients, invasive fungal infection, steroid-sensitive affections (organized pneumonia, non-infectious interstitial involvement, drug-related pulmonary toxicity…), and lung infiltration by the underlying disease (lymphoma, carcinomatous lymphangitis, systemic vasculitis, connective tissue diseases, etc.) were the leading etiologies. No study has evaluated survival benefits from empirical steroids and/or antifungals in immunocompromised patients with ARF from undetermined etiology.

The main objective of this study is to reduce the 90-day mortality in immunocompromised patients with ARF from undetermined etiology at day-3. The intervention would evaluate the impact of steroids ± isavuconazole for 14 days or until ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and < 90 years
* Known immunosuppression:

  1. immunosuppressive drug
  2. solid organ transplant
  3. solid tumor
  4. hematological malignancies
  5. primary immune deficiency
* ICU admission for acute respiratory failure as defined by

  1. respiratory distress with tachypnea (respiratory rate>30/min)
  2. cyanosis
  3. laboured breathing
  4. need for more than 6L of standard oxygen to maintain SpO2>95%, or for high flow oxygen, non-invasive or invasive mechanical ventilation
* No established ARF etiology at day 3
* Informed consent signed:

  * by the patient,
  * Or informed consent signed by a family members/trustworthy person if his condition does not allow him to express his consent in written as per L1111-6,
* Or in an emergency situation and in the absence of family members/trustworthy person, the patient can be enrolled. The consent to participate to the research will be requested as soon as the condition of the patient will allow).

Note: Patient with Pneumocystis pneumonia can be included given that their treatment does not require the use of neither antifungal drugs nor corticosteroids

Exclusion Criteria:

* Patient who improved enough to be discharged from the ICU at day 3
* Documented invasive fungal infection that requires antifungal therapy.
* Patient needing or receiving prophylactic or empirical antifungal treatment for clinical care
* Patient needing or receiving corticoid therapy
* Patient receiving palliative care with comfort measures only (Do Not Intubate (DNI) and Do Not Resuscitate (DNR) patients can be included)
* Pregnant or breastfeeding patient
* No social security coverage
* Known hypersensitivity to isavuconazole or to any of excipients of CRESEMBA® specialty
* Patient treated by ketoconazole, ritonavir, or any CYP3A4/5 inductor
* Short QT syndrome and/or patient with a family history of short QT syndrome;
* Liver insufficiency (any stage)
* Moribund patients
* Participation in another interventional research

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2020-12-21 (Estimated); Primary Completion 2023-09-21 (Estimated); Study Completion 2023-12-21 (Estimated)

PRIMARY OUTCOMES:
Mortality | at day 90
  Overall death

SECONDARY OUTCOMES:
ICU mortality | at ICU discharge within 6 months
  Mortality at ICU discharge
Hospital mortality | at hospital discharge within 6 months
  Mortality at hospital discharge
Mortality | at day 28
  Overall death
Proportion of patients with ICU acquired microbiologically documented bacterial infections | at day 28
Proportion of patients with invasive fungal infection | at day 28
Proportion of patients with herpes simplex virus (HSV) reactivation | at day 28
Proportion of patients with varicella-zoster virus (VZV) reactivation | at day 28
Proportion of patients with cytomegalovirus (CMV) reactivation | at day 28
Occurrence of severe hypokalemia | at day 28
  Severe hypokalemia will be defined as kalemia <2,5 meq/l
Occurence of decompensated diabetes | at day 28
Occurence of severe or newly acquired hypertension | at day 28
Emergence of aspergillus species | at day 28
Incidence of candida infection | at day 28
Incidence of post-traumatic Stress Disorder | at 6 months
  Post-traumatic Stress Disorder will be evaluated using IES-R scale. Impact of Event Scale - Revised (IES-R) is a 22-item self-report measure that assesses subjective distress caused by traumatic events. The higher the score, the more severe the symptoms.
Incidence of anxiety and depression | at 6 months
  Depression and anxiety will be assessed using Hospital Anxiety and Depression Scale (HADS) questionnaire. HADS is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). Limit scores : clearly or clinically symptomatic cases (score ≥ 11).
Quality of life | at 6 months
  Quality of life will be evaluated using SF36. SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting. Items are grouped into three categories: functional status, well-being, overall health assessment. In two dimensions, the answer is binary (yes / no) and in the other 6 in ordinal quality (3 to 6 possible answers). For each dimension, the scores for the different items are coded and then summed and transformed linearly on a scale ranging from 0 to 100. A physical composite score and a mental composite score can be calculated according to an established algorithm

IPD SHARING:
Plan to Share IPD: Undecided